CLINICAL TRIAL: NCT00847925
Title: A Double Blind, Placebo and Standard Care Controlled, Randomised Study to Investigate the Clinical Safety and Toleration, Wound Healing and Antiscarring Potential of Two Applications of Intradermal RN1001 (Avotermin) in Healthy Male Subjects
Brief Title: Safety and Efficacy of RN1001(Avotermin) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: Mark Cooper, Renovo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RN1001-309-1002
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Cicatrix
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- A (Other): 50ng Avotermin/100ul
  Interventions: Drug: Avotermin (RN1001)
- B (Other): 20ng Avotermin/100ul
  Interventions: Drug: Avotermin (RN1001)
- C (Other): 5ng Avotermin/100ul
  Interventions: Drug: Avotermin (RN1001)
- D (Other): 100ng Avotermin/100ul
  Interventions: Drug: Avotermin (RN1001)
- E (Other): 500ng Avotermin/100ul
  Interventions: Drug: Avotermin (RN1001)
- F (Other): 0.25ng Avotermin/100ul
  Interventions: Drug: Avotermin (RN1001)
- G (Other): 1ng Avotermin/100ul
  Interventions: Drug: Avotermin (RN1001)
- H (Other): 20ng Avotermin/100ul
  Interventions: Drug: Avotermin (RN1001)
- I (Other): 50ng Avotermin/100ul
  Interventions: Drug: Avotermin (RN1001)

INTERVENTIONS:
Drug: Avotermin (RN1001) — 100ul/linear cm of wound. Dosed before surgery and 24h later

SUMMARY:
A double blind, Placebo (Vehicle) and Standard Care controlled, randomised study to investigate the clinical safety and toleration (including systemic pharmacokinetics), wound healing and antiscarring potential of two applications of intradermal RN1001 in healthy male subjects

DETAILED DESCRIPTION:
Double blind, randomised, Placebo and Standard Care controlled, single centre study. Each subject served as their own control, i.e. Arm 1 incisions/biopsies randomly received one of two treatments and Arm 2 incisions/biopsies received the same treatments as for Arm 1 but in reverse. The randomisation of the treatment allowed for control of possible positional effects on healing and subsequent scarring. Subjects were initially dosed and wounded (incisions and punch biopsies) on Day 0 and re-dosed on Day 1. On Day 3, Arm 1 incisions and punch biopsies were re-dosed as per Day 0 and excised, and re-dosed again on Day 4. Arm 2 punch biopsies were excised at Day 5 but not re-dosed. Healed incisions/scars on Arm 2 were excised for histological analysis after 12 months and not re-dosed. All subjects, regardless of treatment were treated according to best practices for moist wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-Afro-Caribbean, male subjects aged 18-45 years inclusive.
* Weight between 60 and 150kg and a body mass index between 15 - 55 kg/m2.
* Subjects who have a previous history of surgery or minor injury and who have not developed any evidence of hypertrophic or keloid scar formation

Exclusion Criteria:

* Subjects who on direct questioning and physical examination have history or evidence of hypertrophic or keloid scarring.
* Afro-Caribbean subjects are excluded because of the increased susceptibility to hypertrophic and keloid scarring.
* Subjects with tattoos or previous scars in the areas to be biopsied.
* Subjects, who on direct questioning and physical examination, have evidence of any past or present clinically significant disease and particularly coagulation disorders, immuno mediated conditions and skin diseases and allergies, such as eczema.
* Subjects with a history of clinically significant allergies, especially drug hypersensitivity to lignocaine or allergy to the surgical dressings to be used in this study.
* Subjects with any clinically significant abnormality following review of pre study laboratory data and full physical examination.
* Subjects who are taking, or have taken, certain prescribed or investigational drug in the three weeks prior to Day 0 and in particular topical or systemic steroids, and anti-coagulant drugs. Certain drugs are not excluded in this trial. These include OTC analgesics including paracetamol and codeine, vitamin and mineral supplements, inhaled salbutamol, thyroxine replacement therapy, OTC cold remedies.
* Subjects who drink more than 28 units of alcohol per week (1 unit = ½ pint of beer (285mls) or 25ml of spirits or 1 glass of wine).
* Subjects who have current evidence of drug abuse.
* Subjects who are known to have or had serum hepatitis or who are carriers of the hepatitis B surface antigen or hepatitis C antibody. Subjects with previous vaccination against Hepatitis B are not excluded per se.
* Subjects who are known to have or had serum hepatitis or who are carriers of the hepatitis B core antibody and who show less than 10 units per litre of Anti-HBs.
* Subjects who have previously had a positive result to the test for HIV antibodies, or who admit to belonging to a high-risk group.
* In the opinion of the investigator, a subject who is not likely to complete the study for what ever reason.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2001-11; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Scar severity | 12 Months

SECONDARY OUTCOMES:
Treatment local and systemic tolerance | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Duncan, MB BCh, Principal Investigator — Renovo
Locations (1):
- Renovo CTU, Manchester, United Kingdom

REFERENCES:
- [Derived] Ferguson MW, Duncan J, Bond J, Bush J, Durani P, So K, Taylor L, Chantrey J, Mason T, James G, Laverty H, Occleston NL, Sattar A, Ludlow A, O'Kane S. Prophylactic administration of avotermin for improvement of skin scarring: three double-blind, placebo-controlled, phase I/II studies. Lancet. 2009 Apr 11;373(9671):1264-74. doi: 10.1016/S0140-6736(09)60322-6. PMID 19362676